CLINICAL TRIAL: NCT04705025
Title: Phase II Pilot Study Evaluating the Feasibility of Delivery and Evaluation of a Digital Cognitive-Behavioral Stress Management (CBSM) Device (BNT001) for Treatment of Anxiety and Depressive Symptoms in Patients With Stage I-III Breast or Stage I-III Non-Small Cell Lung Cancer
Brief Title: Cognitive-Behavioral Stress Management Device for the Treatment of Anxiety and Depressive Symptoms in Patients With Stage I-III Breast or Lung Cancer
Acronym: BNT001
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: manufacturer reevaluating Digital cognitive-behavioral stress management (CBSM) device (Attunetm)
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Blue Note Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-002000; NCI-2020-11560 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Lung Non-Small Cell Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
Keywords: Anxiety; depression; cognitive behavioral therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive care (BNT001 app, CBSM, interview) (Experimental): Prior to participating in the study patients complete an online baseline questionnaire to assess anxiety and depression and general quality of life, as well as some specific questions related to their coping. They are also interviewed by a clinician who rates their level of anxiety and depression. After this, patients use the BNT001 app and undergo 10 sessions of CBSM over 45-60 minutes each consisting of cancer-specific educational videos, guided relaxation training, interactive exercises, and discussion modules. Following completion of the 5th session, patients undergo a telephone check-in assessment to see how things are going, update their treatments and medications, and schedule a phone call to assess for adverse events. At the end of the 10th session, patients complete a post-treatment online questionnaire and a phone debriefing interview to discuss their experience with the intervention.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Undergo CBSM using the BNT001 app
  Other Names: CBT; cognitive therapy; CT
Other: Interview — Complete interview
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of a digital application (app), BNT001, on cognitive-behavioral stress management in patients with stage I-III breast or lung cancer. The app is designed for cancer patients to treat anxiety and depressive symptoms related to their cancer diagnosis. The purpose of this study is to develop and refine procedures for eligibility screening, suicide risk assessment, and delivery of the app prior to the launch of a phase III randomized trial. The impact of the app in managing stress and improving quality of life and mood is a secondary aim.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of implementing and evaluating a digital cognitive-behavioral stress management (CBSM) device, BNT001, in stage I-III breast or stage I-III non-small cell lung cancer currently undergoing treatment or recently completed treatment (< 3 months).

SECONDARY OBJECTIVES:

I. To collect preliminary data regarding the efficacy of the intervention with regard to improvements in patients' reported symptoms of distress.

II. To evaluate patient safety and risks associated with screening procedures (severe anxiety or depression) as well as during receipt of the digital intervention.

OUTLINE:

Prior to participating in the study patients complete an online baseline questionnaire to assess anxiety and depression and general quality of life, as well as some specific questions related to their coping. They are also interviewed by a clinician who rates their level of anxiety and depression. After this, patients use the BNT001 app and undergo 10 sessions of CBSM over 45-60 minutes each consisting of cancer-specific educational videos, guided relaxation training, interactive exercises, and discussion modules. Following completion of the 5th session, patients undergo a telephone check-in assessment to see how things are going, update their treatments and medications, and schedule a phone call to assess for adverse events. At the end of the 10th session, patients complete a post-treatment online questionnaire and a phone debriefing interview to discuss their experience with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of stage I-III breast cancer or stage I-III non-small cell lung cancer
* Currently in active treatment or have completed initial cancer directed treatments (surgery, radiation, chemotherapy) within the past 3 months
* Patients showing moderate anxiety (General Anxiety Disorder-7 Questionnaire [GAD-7] > 10) or mild depression (Patient Health Questionnaire depression scale [PHQ-8] score 5-11)
* Fluent in English
* Has access to smartphone or tablet capable of running iOS or Android software

Exclusion Criteria:

* Previous history of cancer
* < 2-year (yr) survival prognosis
* Endorses thoughts of self-harm on question 9 of the Patient Health Questionnaire-9 (PHQ-9) (any score > 0)
* Currently participating in investigative behavioral intervention trial for treatment of anxiety or depression
* Participant is unable to complete training, cognitive deficits, major psychiatric conditions, psycho-social conditions; lack of access to internet accessible device; other social conditions that would interfere with adherence to self-directed care, such that in investigator's opinion the participant would be unable to complete the study
* Recently completed use of Blue Note Therapeutics COVID Cancer Care Program or other Blue Note Therapeutics-sponsored study
* Planning to seek other psychosocial support services while participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing and evaluating the BNT001 digital Cognitive-Behavioral Stress Management device | Up to 1 year
  Feasibility will be evaluated by the rate of recruitment, total number of screens and number of screen fails, treatment adherence (as measured on the backend based on time and regularity of engaging with the digital platform), and number of study completers versus enrolled. The analytic strategy will be primarily descriptive and qualitative. Will also obtain qualitative feedback on participation in the study and study intervention through the end of study de-briefing interview.

SECONDARY OUTCOMES:
Change in global health | Baseline up to 10 weeks
  Change in Patient Reported Outcomes Measurement and Information System (PROMIS)-Global Health Scale v.1.2 using one sample t-tests.
Change in anxiety symptoms | Baseline up to 10 weeks
  Will be assessed by PROMIS-Anxiety version 1.0 using one sample t-tests.
Change in depression symptoms | Baseline up to 10 weeks
  Will be assessed by PROMIS-Depression version 1.0 using one sample t-tests.
Change in anxiety | Baseline up to 10 weeks
  Will be assessed by the Hamilton Rating Scale for Anxiety.
Change in depression | Baseline up to 10 weeks
  Will be assessed by the Hamilton Depression Rating Scale.
Patient safety and risks | Up to 10 weeks
  Will concatenate data regarding the number of individuals requiring severe psychopathology management identified during screening procedures, as well as the number of individuals requiring clinical assessment for severe symptoms during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Ganz, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States